CLINICAL TRIAL: NCT03397771
Title: A Double-Blind Randomised Placebo-Controlled Phase I/IIa Dose Titration Trial to Evaluate the Safety, Tolerability and Efficacy of Oral Litoxetine up to 30 mg vs Placebo BID in Subjects With Urinary Incontinence
Brief Title: DBPC Trial to Evaluate the Safety, Tolerability and Efficacy of Oral Litoxetine in Subjects With Urinary Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ixaltis SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXA-CSP-002
Record Dates: First submitted 2017-12-20; First posted 2018-01-12 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, SSRI
MeSH Terms: conditions — Urinary Incontinence | interventions — litoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind placebo control
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Litoxetine oral capsules (Experimental): oral experimental study medication litoxetine
  Interventions: Drug: Litoxetine
- Placebo oral capsules (Placebo Comparator): oral comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Litoxetine — oral study medication provided in a dose titration manner
  Arms: Litoxetine oral capsules
Drug: placebo — placebo medication provided in a dose titration manner
  Arms: Placebo oral capsules

SUMMARY:
This study will explore the safety, tolerability and efficacy of litoxetine in men and women who suffer from urinary incontinence

DETAILED DESCRIPTION:
This is a double blind randomized placebo controlled study which will explore the safety, tolerability and efficacy of oral litoxetine, a highly selective SSRI, provided by dose titration to subjects suffering from urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

All subjects aged 18 to 70 will be eligible for inclusion in this study if all of the following criteria apply:

1. Willing to provide written informed consent
2. Have symptoms of urinary incontinence for at least 3 consecutive months
3. For male subjects: Undergone prostatectomy at least 6 months prior to inclusion
4. Have at least 7 incontinence episodes per week in the diary entries for the Screening Placebo Run In Period
5. Subject is ambulatory and able to use the toilet independently
6. If subjects use pelvic floor exercises, subjects must have been on a stable exercise and activity regime for at least 3 months prior to screening and that regime must remain stable during the treatment period
7. Subject has a body mass index (BMI) ≥ 19 kg/m2 but ≤ 35 kg/m2 BMI=weight [kg] / height [m2}
8. Subjects must have a pre-dose mean systolic/diastolic blood pressure of ≤ 140/90 mmHg before randomization can occur
9. For female subjects: Must not be pregnant, lactating, or actively trying to become pregnant, Subjects who are premenopausal and of childbearing potential must have a negative pregnancy test at Screening (serum) and at Day 0 (urine) and must use a medically acceptable and effective method of birth control for the duration of the study, which can include:

   1. Having a male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
   2. Use of double-barrier methods of contraception; condoms with the use of caps (with spermicide) and intra-uterine devices are acceptable
   3. Use of hormonal contraceptives (oral, depots, patches, etc.) with double-barrier methods of contraception as outlined above
   4. True abstinence: When this is in line with the preferred and usual lifestyle of the subject (period abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
10. Subjects taking oral contraceptives or hormone replacement therapy (women) or hormone adjuvant therapy (men) must have a stable dose and regimen for ≥ 3 months prior to entry into the study

Exclusion Criteria:

A subject will not be eligible to participate in the study if they meet any of the following criteria:

1. History of anti-incontinence surgery in past 12 months
2. Use of Botox for the treatment of urinary incontinence in the past 12 months
3. Current or recent (3 months) use of any pharmacologic agent used to treat symptoms of urinary incontinence
4. For women: Grade III/IV pelvic organ prolapse; defined per clinical practice
5. For women: History of pelvic prolapse repair or urethral diverticulectomy within 12 months of Screening.

   For men: urethral surgery within 6 months of Screening
6. History of interstitial cystitis or bladder-related pain
7. Subjects with concurrent (at Screening), recent (within 30 days), chronic, or recurrent (> 4 per year) urinary tract infections (positive dipstick for urinary tract infection and abnormal microscopic evaluation, signs and symptoms) or unevaluated microhematuria
8. History of diagnosed gastrointestinal obstructive disorders
9. Chronic severe constipation
10. History of radiation cystitis or history of pelvic irradiation
11. Electrostimulation, biofeedback, or bladder training therapy (behavioural therapy), during the previous month prior to Screening, or the intention to initiate such therapies during the study period. Pessaries and implants are also excluded.
12. Postvoid residual (PVR) urine volume > 150 mL
13. Diagnosis of dementia
14. Diagnosis of epilepsy
15. Diagnosis of acute narrow-angle glaucoma
16. History of mania or diagnosis of bipolar disorder and/or seizures
17. Subjects with uncontrolled hypertension
18. Documented history of myocardial infarction, unstable angina, and/or has undergone coronary artery bypass surgery and/or percutaneous transluminal coronary angioplasty in the past year
19. Congestive heart failure (New York Heart Association Class III or IV heart failure; Appendix 3)
20. Any concurrent condition or any clinically significant abnormality on the Screening physical examination, laboratory tests, electrocardiogram (ECG; including ischemic heart disease), Hepatitis B or C, which, in the opinion of the Investigator, may affect the interpretation of safety or efficacy data, or which otherwise contraindicates participation in a clinical study with litoxetine:

    1. Hypersensitivity to litoxetine or any of its ingredients
    2. History of clinically significant drug hypersensitivity
    3. Subjects with current (within 2 years) urogenital neoplasms or malignancies including bladder, uterine or cervical cancer (not applicable to male subjects with prostate cancer in whom a prostatectomy has been performed)
    4. Subjects with neuropathology that could affect the lower urinary tract or nerve supply, including but not limited to multiple sclerosis, stroke, Parkinsonism, or spinal cord injury
    5. Subjects with diabetes insipidus
    6. Clinically significant or unstable, endocrine, hepatic, renal, immunologic, or lung disease (ie, active chronic obstructive pulmonary disease), or malignancy other than non-melanomatous skin cancer
21. Severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73m2)
22. Severe hepatic impairment (Child-Pugh B or greater)
23. Current or recent (6 months) treatment for depression, or a current diagnosis of depression or have a state of depression or suicidality at Screening.
24. History of current or recent (6 months) suicidal ideation and behaviour (SIB), or history of any suicide attempt in the past 12 months.
25. History of an addiction to drugs or alcohol within 5 years prior to screening, or of alcohol or substance abuse within the past year, as determined by the Investigator. 26. Current use of the following medications:, any serotonergic medication, nonselective irreversible monoamineoxidase inhibitors (MAOIs), cytochrome P450 (CYP)1A2 inhibitors (such as fluvoxamine, ciprofloxacin, or enoxacin), cytochrome P450 (CYP) 2D6 inhibitors (bupropion, fluoxetine, metoclopromide, paroxetine, quinidine), pimozide and thioridazine, and any other medication that would be considered a safety risk for co-administration with litoxetine (See Section 5.7.2 Prohibited Medications)

27. Participation in a clinical study within the month prior to Screening, or exposure to an investigational drug which has not washed out for at least 5 half-lives since its last administration, prior to Screening.

28. In the opinion of the Investigator, is at risk of non-compliance with study procedures, or cannot read, understand, or complete study-related materials (including electronic diaries), particularly informed consent.

29. Participation in any clinical study of an investigational drug that may affect urinary function within 3 months prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Svanberg, Study Director — Ixaltis SA
Locations (1):
- Upstate Clinical Research Associates LLC, Williamsville, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects entered the 2 week Run-in Period and received subject blind placebo treatment. Subjects who continued to meet eligibility criteria at the end of the Run-in Period (at least 7 incontinence episodes per week in the diary entries), entered the Treatment Period, randomly assigned (2:1) to receive study drug (litoxetine) for placebo BID.
Period: Overall Study
Arm/Group | Litoxetine Oral Capsules | Placebo Oral Capsules
Started (Total number is reported as 84; data is reported for 82 subjects as 2 were randomisation errors.) | 53 | 29
Completed | 45 | 22
Not Completed | 8 | 7
Not completed — 2 erroneously randomized, never treated | 3 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: All subjects randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Litoxetine Oral Capsules | Placebo Oral Capsules | Total
Number analyzed (Participants) | 53 | 29 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 23 | 58
  >=65 years | 18 | 6 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 21 | 60
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 38 | 21 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events
Description: AE, SAE, AE of special interest occuring after the start of treatment (LTX or PBP)
Time Frame: from randomisation to treatment completion, an average of 8 weeks
Population: The analysis of TEAE was conducted on the Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Litoxetine Oral Capsules | Placebo Oral Capsules
Number analyzed (Participants) | 53 | 29
Participants | 20 | 10
Statistical Analysis 1: Comparison: Litoxetine Oral Capsules vs Placebo Oral Capsules; Test type: Other; p = 0.963, Regression, Logistic; Odds Ratio (OR) = 1.0

2. Secondary Outcome: Effect Evaluation of Litoxetine for the Treatment of Urinary Incontinence
Description: number of incontinence episodes measured by the use of a bladder diary; change from baseline to week 8 (the higher the number the worse the incontinence severity; minimum value would be zero, there is no limit for maximum value)
Time Frame: change in number of incontinence episodes from baseline to week 8 of treatment
Population: ITT
Measure: Mean (95% Confidence Interval); unit: incontinence events
Arm/Group | Litoxetine Oral Capsules | Placebo Oral Capsules
Number analyzed (Participants) | 46 | 22
incontinence events | -2.05 [-2.57 to -1.54] | -1.20 [-1.81 to -0.58]
Statistical Analysis 1: Comparison: Litoxetine Oral Capsules vs Placebo Oral Capsules; Test type: Non-Inferiority — The analysis was conducted according to the nul hypothesis, assuming no difference between treatment arms; p = 0.022, ANCOVA

ADVERSE EVENTS:
Time Frame: TEAEs were recorded from randomization and through study completion, an average of 8 weeks
Description: The AEs reported refer to TEAEs, ie those AE which occurred after starting randomised treatment and going through week 8 of study.
Arm/Group | Litoxetine Oral Capsules | Placebo Oral Capsules
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/29
Other Adverse Events (participants affected / at risk) | 10/53 | 6/29
OTHER ADVERSE EVENTS (reported when occurring in more than 1.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Litoxetine Oral Capsules (N=53) | Placebo Oral Capsules (N=29)
tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
pyrexia (General disorders) | 1 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
somnolence (Nervous system disorders) | 1 (1) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03397771/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03397771/SAP_001.pdf